CLINICAL TRIAL: NCT02786355
Title: Comparison of Volumes of Air Delivered Through a Frova Intubation Bougie by a Maximal Bimanual Compression Versus a Normal Bimanual Compression of an Adult Ambu® Bag
Brief Title: Oxygenation Via Frova Bougie and Ambu Bag
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Simon Massey, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: H15-03391
Record Dates: First submitted 2016-01-27; First posted 2016-06-01 (Estimated); Results first posted 2018-12-28 (Actual); Last update posted 2018-12-28 (Actual); Status verified 2018-06

CONDITIONS: Failed or Difficult Intubation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maximum bimanual compression (Other): Squeeze through Frova bougie with maximum bimanual compression
  Interventions: Other: Frova bougie
- Normal bimanual compression (Other): Squeeze through Frova bougie with normal bimanual compression
  Interventions: Other: Frova bougie

INTERVENTIONS:
Other: Frova bougie — Squeezing an Ambu bag and delivering air through a Frova bougie. Measuring mean volumes of air delivered and peak pressures generated.

SUMMARY:
We will conduct this study to show that it is possible to deliver air through a Frova bougie and an Ambu® bag.

DETAILED DESCRIPTION:
Participants will be invited to squeeze an Ambu® bag connected to a Frova bougie, and we will measure the volume of air delivered and peak pressure generated.

ELIGIBILITY:
Inclusion Criteria:

* staff, fellows and resident anesthesiologists

Exclusion Criteria:

* injury to hand

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Massey, FRCPC, Principal Investigator — BC Women's Hospital,UBC
Locations (1):
- BC Women's Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dewan P, Taylor J, Gunka V, Albert A, Massey S. Manual volume delivery via Frova Intubating Introducer: a bench research study. Can J Anaesth. 2019 May;66(5):527-531. doi: 10.1007/s12630-019-01308-9. Epub 2019 Feb 12. PMID 30756337

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study design involves a cross-over of participants (i.e., participants are randomly assigned to one of the four groups after which they crossover to the other 3).
Groups:
- Maximum and Normal Effort Using Long and Short Frova Bougies: In a random order, participants would squeeze an Ambu bag attached to a long or short Frova bougie using both maximum and normal effort. As such, participants performed a total of 4 sets of squeezes (maximum effort: long, normal effort: long, maximum effort: short, and normal effort: short) in a random order.
  Frova bougie: Squeezing an Ambu bag attached to a Frova bougie and measuring mean volumes of air delivered.
Period: Overall Study
Arm/Group | Maximum and Normal Effort Using Long and Short Frova Bougies
Started | 35
Completed | 35
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Maximum and Normal Effort Using Long and Short Frova Bougies
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 35

OUTCOME MEASURES:

1. Primary Outcome: Tidal Volume (ml)
Description: volume of air delivered via Frova bougie (milliliters)
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: tidal volume (ml)
Groups:
- Maximum Effort: Long: Squeeze through long Frova bougie with maximum effort
  Frova bougie: Squeezing Ambu bag and ventilating through a Frova bougie and measuring mean volumes of air delivered
- Normal Effort: Long: Squeeze through long Frova bougie with normal effort
  Frova bougie: Squeezing Ambu bag and ventilating through a Frova bougie and measuring mean volumes of air delivered
- Maximum Effort: Short: Squeeze through short Frova bougie with maximum effort
  Frova bougie: Squeezing Ambu bag and ventilating through a Frova bougie and measuring mean volumes of air delivered
- Normal Effort: Short: Squeeze through short Frova bougie with normal effort
  Frova bougie: Squeezing Ambu bag and ventilating through a Frova bougie and measuring mean volumes of air delivered
Arm/Group | Maximum Effort: Long | Normal Effort: Long | Maximum Effort: Short | Normal Effort: Short
Number analyzed (Participants) | 35 | 35 | 35 | 35
tidal volume (ml) | 954.8 (120.7) | 554.4 (131.3) | 893.5 (171.6) | 542.9 (132.9)

ADVERSE EVENTS:
Arm/Group | Maximum and Normal Effort Using Long and Short Frova Bougies
Serious Adverse Events (participants affected / at risk) | 0/35
Other Adverse Events (participants affected / at risk) | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No